CLINICAL TRIAL: NCT06315595
Title: Improvements in Dynamic Contrast-Enhanced MR Angiography and Perfusion and Non-Contrast MRI
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-003511; R01EB031790 (NIH); NCI-2024-01895 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-003511 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Participants undergo a non-contrast MRI on study and may optionally undergo a second non-contrast MRI on study. Participants may also undergo blood sample collection on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates if technical improvements in MRI can be used to provide improved performance contrast-enhanced MRI as used for angiography and perfusion as well as in non-contrast MRI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To study how a variety of technological approaches in MRI can be used to provide improved performance contrast-enhanced MR imaging as used for angiography and perfusion as well as in MR image acquisition without the use of contrast material.

OUTLINE: This is an observational study.

Participants undergo a non-contrast MRI on study and may optionally undergo a second non-contrast MRI on study. Participants may also undergo blood sample collection on study.

ELIGIBILITY:
Inclusion Criteria:

* Adults

Exclusion Criteria:

* Standard exclusion criteria for clinical MRI; e.g. cardiac pacemaker, claustrophobia, an implanted device that has been determined to be MR conditional at 1.5T but not at 3T, anticipated considerable susceptibility artifact from hip prosthesis, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult male volunteers as well as Mayo patients for whom a prostate MRI exam has been clinically indicated and ordered. In some cases such as for evaluation of the vasculature of the pelvis it may be useful to extend the inclusion criteria of volunteers to adult females.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09-30 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Improved performance in contrast-enhanced magnetic resonance imaging (MRI) as used for angiography and perfusion | Baseline (at enrollment); possible second scan at a later date
  Assessed by comparison of two images made from the raw data set but reconstructed using the standard vs. an alternative algorithm (to be determined during study). Data will be tabulated and analyzed statistically.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Riederer, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials